CLINICAL TRIAL: NCT00417885
Title: Phase 1/2 Open-Label Trial Of Sutent (Sunitinib Malate) And Aromasin(Exemestane) In The First-Line Treatment Of Hormone Receptor-Positive Metastatic Breast Cancer
Brief Title: A Clinical Trial Assessing Efficacy and Safety of Sunitinib and Exemestane in Patients With ER [Estrogen Receptor] + and/or PgR [Progesterone Receptor] + Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: See Detailed Description for Termination Reason
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181108
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): sunitinib + exemestane
  Interventions: Drug: exemestane; Drug: sunitinib malate

INTERVENTIONS:
Drug: exemestane — 25 mg, oral, daily dosing
Drug: sunitinib malate — 37.5 mg, oral, continuous dosing, daily
  Other Names: sutent

SUMMARY:
To assess progression-free survival at the combination dose determined in the Phase 1 portion of the study, and safety of sunitinib combined with exemestane in patients with metastatic or locally-recurrent, unresectable breast cancer.

DETAILED DESCRIPTION:
The trial was terminated prematurely on August 28, 2008 due to the inability to recruit the planned number of subjects in order to provide meaningful efficacy data. There were no safety concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Estrogen and/or progesterone receptor positive adenocarcinoma of the breast with evidence of 1) unresectable 2)locally recurrent, or 3) metastatic disease
* Postmenopausal
* ECOG [Eastern Cooperative Oncology Group] </=1
* Evaluable(e.g bone only disease allowed) and Measurable disease [RECIST (Response Evaluation Criterion in Solid Tumors)]

Exclusion Criteria:

* HER2 [Human Epidermal Growth factor Receptor 2] positive disease not previously treated with herceptin
* Any prior anti-angiogenic therapy, endocrine or cytotoxic anti-cancer therapy in the metastatic disease setting
* Radiation therapy within 2 weeks of first study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Atlanta, Georgia, United States
- Pfizer Investigational Site, Montreal, Quebec, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181108&StudyName=A%20Clinical%20Trial%20Assessing%20Efficacy%20and%20Safety%20of%20sunitinib%20and%20exemestane%20in%20Patients%20with%20ER+%20and/or%20PgR+%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + Exemestane: Sunitinib administered orally, in a continuous regimen, dose of 37.5 mg daily. Exemestane coadministered orally at a dose of 25 mg daily.
Period: Overall Study
Arm/Group | Sunitinib + Exemestane
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Objective Progression or Relapse | 3
Not completed — Transferred to Another Sunitinib Study | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  < 18 years | 0
  18 to 44 years | 0
  45 to 64 years | 4
  > = 65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from enrollment to first documentation of objective tumor progression or to death on study due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. PFS was to be calculated as (first event date - the date of enrollment +1)/7.
Time Frame: From start of treatment until Day 1 of every other cycle (8 weeks) or death
Population: Intent-To-Treat (ITT) = all subjects who were enrolled in the trial. Data were not analyzed due to early termination.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response (OR) According to the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: OR=from start of treatment until disease progression/recurrence. Complete response (CR)=disappearance of all target lesions. Partial response (PR)= ? 30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions. Progressive disease (PD)= ? 20% increase in sum of longest dimensions of lesions taking as reference smallest sum of the longest dimensions since treatment started, or appearance of ? 1 new lesion. Stable disease (SD)=neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: From start of treatment until Day 1 of every other cycle (8 weeks)
Population: Analyses on OR were performed for subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 6
participants
  CR | 1
  PR | 1
  PD | 1
  SD | 3

3. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death on study. If tumor progression data included more than 1 date, the first date was used. DR was to be calculated as (the end date for DR - first CR or PR that was subsequently confirmed +1)/7.
Time Frame: From start of treatment until Day 1 of every other cycle (8 weeks) or death due to cancer
Population: Analyses on DR were to be performed for overall responders only. Data were not analyzed due to early termination.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of enrollment to date of death due to any cause. OS was to be calculated as (the event date - the date of enrollment +1)/7.
Time Frame: From start of study treatment until death
Population: ITT. Data were not analyzed due to early termination.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from enrollment to first documentation of objective tumor progression. If tumor progression data included more than 1 date, the first date was used. TTP was to be calculated as (first event date - the date of enrollment +1)/7.
Time Frame: From start of treatment until Day 1 of every other cycle (8 weeks)
Population: ITT. Data were not analyzed due to early termination.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 0

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The clinical benefit rate (CBR) was the measure for clinical benefit (CB) and was defined as the percent of subjects with confirmed CR or confirmed PR, or confirmed SD according to RECIST, relative to the total analysis population. CRs were those that persisted on repeat imaging study ?4 weeks after initial documentation of response.
Time Frame: From start of treatment until Day 1 of every other cycle (8 weeks)
Population: ITT. Data were not analyzed due to early termination.
Measure: Number; unit: rate
Arm/Group | Sunitinib + Exemestane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sunitinib + Exemestane
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Exemestane (N=6)
Pancreatitis acute (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Enterobacter sepsis (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Exemestane (N=6)
Leukopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Diabetes insipidus (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Diplopia (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Myodesopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 1
Fatigue (General disorders) | 5
Fibrosis (General disorders) | 1
Induration (General disorders) | 1
Influenza like illness (General disorders) | 1
Irritability (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Weight decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Micturition urgency (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Vaginal disorder (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.